CLINICAL TRIAL: NCT05885490
Title: Protocol for The International Centre for Recurrent Head and Neck Cancer (IReC) Tissue Biobank and Data Registry
Brief Title: IReC-Bio and IReC Registry
Acronym: IReC-Bio
Status: Not yet recruiting | Type: Observational
Sponsor: Royal Marsden NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: 5604
Record Dates: First submitted 2023-05-03; First posted 2023-06-02 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Head Cancer Neck
MeSH Terms: conditions — Head and Neck Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Surplus tumour tissue and an optional EDTA blood sample will be collected
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Group 1: Patients undergoing treatment for histologically proven or suspected recurrent cancer of the head and neck - clinical data only
- Group 2: Patients undergoing treatment for histologically proven or suspected recurrent cancer of the head and neck - clinical data and optional biobank sampling
- Group 3: Patients undergoing treatment for histologically proven or suspected recurrent cancer of the head and neck - clinical data and optional quality of life data
- Group 4: Patients undergoing treatment for histologically proven or suspected recurrent cancer of the head and neck - clinical data and optional quality of life data and optional biobank sampling

SUMMARY:
IReC is the world's first centre for recurrent head and neck cancers. We have the ambitious aim to create a centre of international excellence and set international standards in the curative treatment of recurrent head and neck cancers.

One of IReC's key objectives is to develop a national research tissue bank to support laboratory and translational research. The cornerstone of translational research is a well-annotated biobank of cancer samples to explore and validate key research findings.

The purpose of IReC-Bio is to support research into recurrent head and neck cancers. A central repository for the rarer recurrent cancers will allow the concentration of cases required in order to support translational research programmes. The overall aim is to facilitate research into understanding disease biology, identifying potentially curative treatments, and allow detailed investigations into the relationships between clinical, pathological and molecular characteristics and clinical outcomes.

Combining the IReC Registry and Biobank gives us a comprehensive data and sample set which has never been created before for recurrent head and neck cancer. The aim is to have a national, and in the future international, resource of the study of recurrent head and neck cancer on a molecular and clinical level to support novel ways of treating rHNC.

DETAILED DESCRIPTION:
There are currently only a limited number of proven treatments for use in cancers of the head and neck, and a better understanding of the biology of different HNCs could lead to improved therapies. Although many patients with head and neck cancer can be offered potentially curative treatment, we do not understand why some people are cured and others are not. There has been an explosion in molecular research in many cancers, but this remains an understudied area in head and neck cancer. There are currently no treatments available to patients with head and neck cancer based on molecular characteristics.

The purpose of IReC-BIO is to support research into rHNCs. A central repository for the rarer recurrent cancers will allow the concentration of cases required in order to support translational research programmes. The overall aim is to facilitate research into understanding disease biology, identifying potentially curative treatments, and allow detailed investigations into the relationships between clinical, pathological and molecular characteristics and clinical outcomes.

Cancer registries store large quantities of data from defined cancer populations. Registry aims vary, but include analysing cancer trends over time and supplying data for research studies5-7. The NCDB and SEER are extensively studied registries, producing >200 publications per year6. Both provide a broad overview of all major cancers; however, they have notable datapoint gaps, in particular, recurrence and patient reported outcome measures (PROMs).

Establishing a cancer registry necessitates a balance of clinical, informatic, and financial influences. Cancer registry development is subject to numerous pitfalls, ranging from excessive datapoints to inadequate quality assurance7. These can be mitigated through adherence to best practice recommendations, for example the NAACCR and ENCR, which provide guidelines that standardise registry datasets8,9. However, not all recommendations are practical across all cancer diagnoses. In particular, rHNC requires a tailored approach to document the treatment and functional implications unique to this cohort, necessitating development of a registry specific to this disease.

ELIGIBILITY:
Inclusion Criteria:

* Aged over 18 at time of diagnosis.
* Confirmed clinical, radiological, and/ or histological diagnosis of residual, recurrent, or new primary malignant head and neck cancer arising from the nasopharynx, oropharynx, oral cavity, larynx, hypopharynx, sinonasal cavities, major salivary glands and thyroid gland.
* Any mucosal, salivary gland, and thyroid histological subtype
* Ability to give informed consent.
* Details of clinical follow-up available

For IReC-BIO only:

* FFPE blocks(s) or fresh frozen tumour tissue available for collection
* Two or more tumour-containing blocks available from the same specimen

For QoL Questionnaires only:

• Patients who have received a diagnosis of rHNC no earlier than 6 weeks prior to study entry

Exclusion Criteria:

• Recurrent cutaneous (e.g., SCC, melanoma), sarcomatous, and lymphatic or haematological (e.g. lymphoma) malignancies of the head and neck

For IReC-BIO only:

* FFPE tumour samples contain insufficient tumour sample for analysis.
* Insufficient clinical details available

For QoL Questionnaires only:

• Patients who have received a diagnosis of rHNC more than 6 weeks prior to study entry

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients undergoing treatment for histologically proven or suspected recurrent cancer of the head and neck
Sampling Method: Probability Sample
Enrollment: 10000000 (Estimated)
Dates: Start 2026-04 (Estimated); Primary Completion 2050-12 (Estimated); Study Completion 2050-12 (Estimated)

PRIMARY OUTCOMES:
Define the 2 year overall survival rates in all patients with rHNC | 2 years
  2-year overall survival from date of diagnosis

SECONDARY OUTCOMES:
Define the 2-year disease-free (DFS), disease-specific (DSS), and local recurrence free survival (LRFS) rates in all patients with rHNC. | 2 years
  2 year disease free survival, disease specific and local recurrence free survival rates in all patients with rHNC
Define long-term functional outcomes after diagnosis of rHNC using gastrostomy and tracheostomy use as a surrogate marker up to 2 years after diagnosis with rHNC | 2 years
  1 and 2-year gastrostomy and tracheostomy status from date of diagnosis
Assess swallow with Performance Status Scale for head and neck cancer patients (PSS-HN) scores up to 2 years after diagnosis of rHNC. | 2 years
  Entry, 6, 12 and 24-month PSS-HN NOD scores